CLINICAL TRIAL: NCT01842347
Title: Treatment of C. Difficile Infection With Fecal Microbiota Transplantation (FMT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Steve Werlin, MD, Professor, Principal Investigator, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pediatrics, C. Diff. (Experimental): Fecal Microbiota Transplantation in children with c. difficile infection
  Interventions: Other: Fecal microbiota

INTERVENTIONS:
Other: Fecal microbiota

SUMMARY:
The purpose of this study is to treat children with severe, moderate, resistant or relapsing C. difficile infection and to determine the changes in the intestinal microbiome (all of the bacteria living in the intestines) in children receiving FMT for C. difficile infection. Data will be collected throughout the FMT procedure to determine effectiveness and to help standardize this procedure. Stool samples will be collected to look at the different bacteria that are in the intestines before and after FMT.

ELIGIBILITY:
Recipient Inclusion Criteria

1. Older than 18 months of age
2. FMT procedure has been decided by the treating gastroenterologist and was based on:

   1. Recurrent or relapsing CDI and:

      * Failure of standard medical therapy with metronidazole, vancomycin and fidaxomicin (over age 18 years. Fidaxomicin is not approved for <18years and insurance authorization may not be possible).
      * At least 2 episodes of CDI requiring hospitalization
   2. Moderate CDI not responding to vancomycin for at least a week.
   3. Severe CDI with no response to vancomycin after 4 hours.
3. English speaking

Recipient Exclusion Criteria

1. Lack of informed consent/assent.
2. Not eligible for FMT procedure

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Treatment of C. Difficile Infection with Fecal Microbiota Transplantation (FMT) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Werlin, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States